CLINICAL TRIAL: NCT01202708
Title: Safety and Efficacy of Hemodiafiltration With On-Line Preparation of Substitution Fluid Using the Gambro AK 200 ULTRA System
Brief Title: Gambro AK200 ULTRA Hemodiafiltration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 070003
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Renal Failure
Keywords: chronic renal failure; hemodiafiltration
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: On line hemofiafiltration — hemodiafiltration with the Gambro AK 200 ULTRA
  Other Names: Gambro AK 200 ULTRA
Device: On line hemodiafiltration — On line hemodiafiltration with the Gambro AK 200 ULTRA System
  Other Names: Gambro AK 200 ULTRA System

SUMMARY:
This study is designed to assess the safety, efficacy and dialytic capabilities of hemodiafiltration with on-line prepared substitution fluid using the AK200 ULTRA in comparison to conventional hemodialysis.

DETAILED DESCRIPTION:
The AK200 ULTRA is a new device in the United States, but has been used for several years in Europe. The AK200 ULTRA is a single unit which is preprogrammed to provide standard hemodialysis as well as hemofiltration and hemodiafiltration with on-line preparation of the substitution fluid The AK200 ULTRA hemofiltration and hemodiafiltration is performed using a high flux membrane with high ultrafiltration rates compensated by volumetrically controlled infusion of on-line prepared substitution fluid. The AK200 ULTRA is, therefore, capable of providing dialysis treatments which can improve the removal of medium to high weight molecules without the difficulties associated with the manual measurement and administration of external substitution fluid.

This study is designed to assess the safety, efficacy and dialytic capabilities of hemodiafiltration with on-line prepared substitution fluid using the AK200 ULTRA in comparison to conventional hemodialysis. This study is motivated by the need for a commercially available product capable of administering hemofiltration and hemodiafiltration in a clinical setting. The ultimate goal of this study is to improve morbidity and mortality in the ESRD patient population in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Subject received chronic dialysis therapy
2. Subject was stable on three dialysis sessions per week
3. Subject was able to understand and sign the informed consent

Exclusion Criteria:

) On chronic renal replacement therapy for less than three (3) months 2) Hospitalization for reasons other than vascular access complications in the past three (3) months 3) HIV + 4) Hepatitis B+ 5) Pregnancy, verified by pregnancy test for women of child bearing potential 6) Access recirculation > 10% 7) Hematocrit less than 26% 8) History of non compliance 9) Pediatric patients, defined as less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1997-08; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Primary Goal: To assess the safety and efficacy of hemodiafiltration with on-line prepared substitution fluid using the AK200 ULTRA for the treatment of chronic renal failure. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Susie Q. Lew, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Center, Washington D.C., District of Columbia, United States